CLINICAL TRIAL: NCT05479669
Title: Value of Intense Phenotyping in Heart Failure With Preserved Ejection Fraction
Acronym: VIP-HF2
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: VIP-HF 2
Record Dates: First submitted 2022-07-19; First posted 2022-07-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure, Diastolic
Keywords: heart failure with preserved ejection fraction; HFpEF; cardiac MRI; 99mTc-HDP scan
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Echocardiography; Electrocardiography, Ambulatory; Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — Transthoracic echocardiograms will be performed at inclusion. Echocardiographic parameters that will be evaluated are measures of atrial size (including left atrial volume, right atrial dimensions, left ventricular function and dimensions (including left ventricular dimensions, septal wall thickness, posterior wall thickness, systolic function, Simpson biplane left ventricular ejection fraction), parameters of diastolic dysfunction (including E, A, E/A ratio, deceleration time, E' and E/E' ratio) and valve (dys)function.
Diagnostic Test: 24 hour Holter monitoring — 24-hours Holter monitoring will be used to determine markers of increased risk of ventricular arrhythmias, such as non-sustained ventricular tachycardias, and ventricular premature beats and doublets. Also the presence and pattern of AF and runs of supraventricular tachycardias are determined.
Diagnostic Test: Cardiac Magnetic Resonance Imaging — Multiple short-axis cine images will be acquired throughout the entire LV with a steady-state free precession sequence. Left ventricular volumes, ejection fraction and myocardial mass will be measured on the short-axis stacks at end diastolic and end systolic frames. Ten to 15 minutes after an intravenous bolus injection of a gadolinium-based contrast agent late gadolinium enhancement will be performed with a segmented inversion recovery gradient-echo sequence, using the same image orientation as in the short-axis stacks. The presence, location and morphology of myocardial fibrosis will be described. The extent of myocardial scar will be quantified using computer-assisted planimetry and expressed as a percentage of left ventricular mass. Pre- and post-contrast T1 measurements will be obtained using a single-shot modified Look Locker inversion recovery sequence. Extracellular volume (a measure of diffuse myocardial fibrosis) will be quantified.
Diagnostic Test: 99mTc-HDP scan — Patients will receive a 99mTc-HDP scan. 3 hours after the technetium 99m-hydroxymethylene diphosphonate bolus injection, imaging will be performed using a gamma-camera equipped with a collimator which guides individual gamma-rays emitted by the radionuclide. For planar imaging, a collimator will be used to transfer only those gamma-rays which pas in a perpendicular course. Sequentially, a SPECT-CT will be performed in the same session to improve sensitivity. SPECT/CT will be performed on a SPECT/CT dual head gamma camera system. SPECT images will be acquired using a 128 x 128 matrix, 180 degrees of rotation, 64 views, 15s per view. Visual image analysis will be performed by two blinded and experienced nuclear medicine physicians. Data will be scored according to a routine scoring system on a scale from 0 (no cardiac uptake of 99m technetium and normal bone uptake) to 3 (high cardiac uptake, higher than bone uptake).
Diagnostic Test: ECG — A 12-lead electrocardiogram will be performed at the 1-year and 2-year follow-up visit to determine the heart rhythm and heart rate.

SUMMARY:
Heart failure (HF) with a left ventricular ejection fraction (LVEF) >0.40 is a large medical problem, for which no drug or device has a recommendation in current HF guidelines. The prevalence of mortality and HF hospitalizations in HF with LVEF >0.40 is high, but the identification of predictors for increased risk of mortality and HF hospitalizations in this patient category remains difficult. The hypothesis of this study is that the risk of all-cause mortality and HF hospitalizations can be measured by clinical factors, imaging parameters and circulating biomarkers, and that these factors can be used in a risk profile

DETAILED DESCRIPTION:
Objective: To assess the risk profile associated with the combined endpoint of all-cause mortality and HF hospitalizations in HF patients with LVEF >0.40.

Study design: Single-center, prospective, study.

Study population: We aim 200 patients with symptomatic heart failure (NYHA class II-III), and a recent HF hospitalization, emergency room visit or symptom relief with diuretics who have a left ventricular ejection fraction >0.40, echocardiographic evidence of left atrial enlargement or left ventricular hypertrophy, and elevated concentrations of BNP or NT-proBNP.

Study procedures: All patients will undergo echocardiography, cardiac magnetic resonance (CMR) imaging, Holter recording and blood sampling at inclusion. The 99mTc-HDP scan is optional.There is no control group.

Total follow up: Up to five years.

Main study endpoint: incidence of the combined endpoint of all-cause mortality and HF hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

Clinical criteria:

1. Age >18 years
2. Written informed consent
3. HF with moderate to severe symptoms NYHA II or III
4. Hospitalization or emergency room visit for HF or symptom relief with diuretics
5. Sinus rhythm or AF

Echocardiographic criteria:

1. LVEF >0.40
2. Left atrial size (volume ≥29 mL/m2 or LA parasternal diameter ≥45), or left ventricular hypertrophy (septal thickness or posterior wall thickness ≥11 mm) or LV diastolic dysfunction (E/e' ≥13 or mean e' septal and lateral wall <9 cm/s).

Biomarker criteria:

1. BNP >31ng/L or NT-pro-BNP>125ng/L if sinus rhythm
2. BNP >75ng/L or NT-pro-BNP>300ng/L if atrial fibrillation

Exclusion Criteria:

1. Patients unwilling or unable to sign informed consent
2. Patients with a pacemaker or ICD
3. Indication for ICD therapy according to the ESC guidelines
4. Life expectancy of less than one year
5. Significant coronary artery disease or myocardial infarction < 3 months
6. Complex congenital heart disease
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To avoid the inclusion of patients with dyspnea due to other causes, we use specific (see below) echocardiographic and biomarker criteria. From several studies is known that in patients with HF with LVEF >0.40 or AF, NT-proBNP or BNP is strongly associated with mortality an HF hospitalizations. The use of biomarker criteria will therefore help to select patients with an increased mortality risk. Therefore, by selecting HF patients with LVEF >0.40 with a previous HF hospitalization we aim to include patients at increased risk for mortality and HF hospitalizations.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint of all-cause mortality and hospitalization for heart failure | 5 years
  The incidence of the combined endpoint of all-cause mortality and first heart failure hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Rienstra, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No